CLINICAL TRIAL: NCT04604093
Title: Use of the FreeStyle Libre 2 Flash Glucose Monitoring System to Reduce Hyperglycemia in People With T2 Diabetes
Brief Title: Effect of the FreeStyle Libre 2 Flash Glucose Monitoring System on Hyperglycemia in People With T2 Diabetes
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-20193
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SMBG, self-monitoring of blood glucose: Subjects will be randomized to continue use traditional SMBG, self-monitoring of blood glucose, to manage their diabetes.
  Interventions: Device: SMBG Meter
- FreeStyle Libre 2: Subjects will be randomized to use the FreeStyle Libre 2 Flash Glucose Monitoring System to manage their diabetes.
  Interventions: Device: FreeStyle Libre 2 System

INTERVENTIONS:
Device: SMBG Meter — Self Monitoring Blood Glucose Meter
  Groups: SMBG, self-monitoring of blood glucose
Device: FreeStyle Libre 2 System — The Abbott's FreeStyle Libre 2 Flash Glucose Monitoring System
  Groups: FreeStyle Libre 2

SUMMARY:
A multi-center, randomized, prospective, non-significant risk study to compare the impact of the FreeStyle Libre 2 Flash Glucose Monitoring System to the current standard of care (SMBG, self-monitoring of blood glucose) on reducing time above 180 mg/dL in subjects with type 2 diabetes who are not adequately controlled on their existing oral anti-diabetes medication regimen.

DETAILED DESCRIPTION:
Up to approximately 350 subjects will be enrolled to obtain a minimum of 130 randomized subjects, with a minimum of approximately 65 subjects per arm. At least 50% of randomized subjects will be age 65 and older. Subjects will be randomized to use either the FreeStyle Libre 2 Flash Glucose Monitoring System or traditional SMBG to manage their diabetes. The subsequent impact of FreeStyle Libre 2 versus SMBG on reducing the amount of time spent above 180 mg/dL will be assessed.

Safety of the FreeStyle Libre 2 Flash Glucose Monitoring System and SMBG will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have HbA1c of > 7.5% at screening
3. Subject has 35% or more time spent above 180 mg/dL during the screening phase.
4. Subject must have had a diagnosis of type 2 diabetes for at least six (6) months prior to enrollment.
5. Subject has been prescribed at least one capillary blood test every day for self-management of blood glucose (SMBG) to manage their diabetes.
6. Subject must be on at least one (1) oral anti-diabetes medication.
7. Subject must be able to read and understand English.
8. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
9. Subject is willing to make diet and lifestyle changes in response to education and glucose data
10. Subject must be available to participate in all study visits.
11. Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

1. Subject is currently on any form of insulin therapy.
2. Subject has used an unblinded continuous glucose monitor (CGM) in the 3 months prior to enrollment.
3. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
4. Subject is known to be pregnant at the time of study enrollment (applicable to female subjects only).
5. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
6. Subject has concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
7. Subject is currently undergoing dialysis and/or has end stage renal disease.
8. Subject is currently participating in another interventional clinical trial.
9. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with type 2 diabetes diagnosis currently on oral anti-diabetes medication(s).
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Impact on time above 180 mg/dL in subjects with type 2 diabetes | Six (6) months
  To assess the impact of the FreeStyle Libre 2 Flash Glucose Monitoring System on time above 180 mg/dL in subjects with type 2 diabetes who are not adequately controlled on their existing oral anti-diabetes medication regimen when compared to the current standard of care (SMBG, self-monitoring of blood glucose).

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care Inc
Locations (5):
- United States (5):
  - Valley Research, Fresno, California
  - CEDE (Center of Excellence in Diabetes and Endocrinology), Sacramento, California
  - Metabolic Research Institute, West Palm Beach, Florida
  - Billings Clinic, Billings, Montana
  - Palm Research Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No